CLINICAL TRIAL: NCT04714112
Title: Comparison of the Effects of Different Time of Intravenous Dexamethasone on Brachial Plexus Block: a Randomized Control Study
Brief Title: Low-dose Intravenous Dexamethasone at Different Times as Adjunvants for Brachial Plexus Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Quanhong Zhou, Principal Investigator, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-186
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Analgesia; Dexamethasone; Brachial Plexus Block; Intravenous Drug Usage; Time; Shoulder Surgery
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative group (Experimental): Intravenous dexamethasone (5mg) is used when ultrasound guided ISB is performed.
  Interventions: Drug: dexamethasone
- postoperative group (Active Comparator): Ultasound guided ISB is performed before operation and intravenous dexamethasone (5mg) is used in postoperative care unit ( PACU)
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — Intravenous administration of dexamethasone at different time for the duration of ISB with 0.5% ropivacaine
  Other Names: Dexamethasone Dexamethasone sodium phosphate

SUMMARY:
Dexamethasone has been tested as an effective adjuvant to prolong the effect of local anesthetics for peripheral nerve blocks, both perineurally and intravenously. The purpose of this study is to investigate the effect of the addition of dexamethasone (5mg) at different time to a standard ropivacaine solution (0.5%) on analgesic duration of interscalene block.

DETAILED DESCRIPTION:
Interscalene brachial plexus block (ISB) is regarded as the standard of care for anesthesia and analgesia for shoulder surgery by providing the superior analgesia and reducing opioid consumption. After several hours when the effects of single injection ISB wear off, the patients often suffer moderate to severe pain of the surgical insult and required strong opioid analgesia. Efforts to prolong ISB duration by adding adjuvants to local anesthetic (eg. clonidine, dexmedetomidine) have been studied with promising results. Dexamethasone, has been added to local anesthetic solutions for ISB and has demonstrated promise in preliminary studies. Perineural dexamethasone (8-10mg) in conjunction with local anesthetic prolongs the duration of ISB with an effect sizes ranging from 40% to 75% (absolute effect ~ 6 to 10 hours). Dexamethasone, however, is only approved for intramuscular or intravenous administration and therefore perineural use is currently off-label. Intravenous administration of dexamethasone was reported to have similar effects as perineural route indicating the possible mechanism for prolonging analgesic duration might be due to the systemic effects of dexamethasone. We hypothesized: should that is the reason, systemic administration of dexamethasone at different time may provide similar effects on the duration of peripheral nerve block. Dexamethasone is a slow effect cortisone with long half-time, it is widely used at the beginning of surgery to prevent postoperative nausea and vomiting. A trial that demonstrates enhanced block quality and duration associated with intravenous dexamethasone at different time may allow us to achieve prolonged duration of effect if dexamethasone is used in perioperative period for different purpose. This would further identify the possible mechanism of dexamethasone to prolong the analgesia effect of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic shoulder surgery at Shanghai Sixth People's Hospital.
* ASA functional status class I to II
* Age 18 to 70 years
* BMI ≤ 35 kg/m2

Exclusion Criteria:

1. Lack of patient consent
2. Allergy to dexamethasone or ropivacaine
3. BMI > 35 kg/m2
4. Contraindications to low dose dexamethasone including peptic ulcer disease, systemic infection, glaucoma, active varicella/herpetic infections, diabetes mellitus
5. Contraindications to ISB including severe Chronic Obstructive Pulmonary Disease (Forced expiratory volume < 40% predicted), coagulopathy, pre-existing neurologic deficit in ipsilateral upper extremity, localized infection
6. Pregnant or nursing females
7. Chronic opioid use defined as > 30mg oral morphine or equivalent per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | one day postoperative
  from completion of ISB to VAS for pain > 0 ( in hours)

SECONDARY OUTCOMES:
Time to First Opioid Consumption | one day postoperative
  Time from completion of block procedure to first consumption of opioid analgesic (in hours)
Opioid Consumption | two days postoperative
  Opioid consumption (in oral morphine equivalents) will be recorded at 12 hours, 24 hours and 48 hours
Visual Analog Scale for pain ( from 0 to 10 ) | 7 days postoperative
  Recorded at 12 hours, 24 hours, and 7 days 0 is no pain, 10 is the worst pain imaginable. Lower number is better.
Postoperative Serum Blood Glucose | one day postoperative
  Measured on the morning of first day after surgery
Infection | 7 days postoperative
  Number of participants with localized infection at nerve block site
Number of Participants With Postoperative Nausea and/or Vomiting | 7 days postoperative
  Number of participants with postoperative nausea and/or vomiting assessed at 12 hours, 24, hours, and 7 days postoperatively
Number of Participants With Nerve Damage From Interscalene Block | 7 days postoperative
  Persistent paresthesia, and sensory/motor block at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Quanhong Zhou, MD., Ph.D, Principal Investigator — Shanghai Jiaotong University affiliated Shanghai Sixth People's Hospital
Locations (1):
- Shanghai Jiaotong University affiliated Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No